CLINICAL TRIAL: NCT03466996
Title: Telemedicine in Spina Bifida Transition: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's of Alabama (Other)
Responsible Party: Principal Investigator, Elizabeth Kuhn, Principle Inverstigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-555555
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Spina Bifida
Keywords: Transition to adult care; Telemedicine; Myelomeningocele
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in face-to-face video telemedicine visits, in addition to routine annual visits to the Spina Bifida Clinic. These 30-minute visits will occur at 2 weeks, 3 months, 6 months and 9 months from last in-person clinic appointment. The visits will consist of structured counseling using a plan-do-study-act cycle approach to incrementally adopt elements of a well-planned transition. Using qualitative notes from each session, we will identify common themes or challenges across patients and develop adjunctive education, support, and monitoring tools for patients and families in transition.
  Interventions: Behavioral: Intervention group
- Standard of care group (Active Comparator): The control group will receive the current standard of care transition program. In addition to this, they will receive encouraging text messages and e-mails relating to their transition goals. These messages will be sent 2 weeks, 3 months, 6 months and 9 months from the last in-person clinic appointment.
  Interventions: Behavioral: Standard of care group

INTERVENTIONS:
Behavioral: Intervention group — More frequent follow up with face to face interaction.
  Other Names: Telemedicine group
  Arms: Intervention group
Behavioral: Standard of care group — Transition goal setting during annual follow up.
  Arms: Standard of care group

SUMMARY:
The purpose of this study is to explore the feasibility and efficacy of using telemedicine to improve transition from pediatric to adult care in patients with spina bifida.

DETAILED DESCRIPTION:
After enrollment, patients will be randomly assigned to either the control or intervention group. Randomization will be performed using computer software with 1:1 group allocation. We anticipate 26 participants in each group.

The control group will receive the current standard of care transition program which includes goal-setting at their annual Multidisciplinary Spina Bifida Clinic visit. Additionally, they will receive encouragement e-mail and text messages. These messages will be sent at 2 weeks, 3 months, 6 months, and 9 months from last in-person appointment.

The intervention group will participate in face-to-face video telemedicine visits, in addition to routine yearly visits to the Spina Bifida Clinic. These 30-minute visits will occur at 2 weeks, 3 months, 6 months and 9 months from last in-person clinic appointment. The visits will consist of structured counseling using a plan-do-study-act cycle approach to incrementally adopt elements of a well-planned transition. Using qualitative notes from each session, I hypothesize that I will be able to identify common themes or challenges across patients and develop adjunctive education, support, and monitoring tools for patients and families in transition. I will collaborate with experts from orthopedic surgery, physical medicine and rehabilitation, urology, neurosurgery, nutrition, and psychology to develop content for educational tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 13 years with a diagnosis of spina bifida who are currently seen through the Children's of Alabama Multidisciplinary Spina Bifida Clinic

Exclusion Criteria:

* Patients without access to the internet.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Transition preparedness | Baseline to 12 months
  Transition preparedness will be assessed using Transition Readiness Assessment Questionnaire (TRAQ), a validated, patient-centered questionnaire. Each item is scored 1-5, with 1 being assigned for responses of "No, I do not know how"(not ready for transition) and a score of 5 assigned for responses of "Yes, I always do this when I need to."(ready for transition).
Health-related quality of life | Baseline to 12 months
  Health-related quality of life (HRQoL) will be assessed using the generic Pediatric Quality of Life InventoryTM (PedsQLTM). 0-100 scale, the higher scores indicate better quality of life.
Improvement in bowel management | Baseline to 12 months
  Spina bifida-specific Quality of Life Assessment in Spina Bifida for Children (QUALAS-C) (a measure of bowel and bladder-related HRQoL). QUALAS-T is scored 0-100, where higher values signify higher HRQOL.

SECONDARY OUTCOMES:
Healthcare utilization | Baseline to 24 months
  Number of hospitalizations; ER and clinic visits.
Health care related cost | Baseline to 24 months
  We will track number of hospitalizations, ER and clinic visits as related to cost. The goal is to reduce these visits.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kuhn, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States